CLINICAL TRIAL: NCT02589262
Title: A Randomised, Double-blind, Placebo-controlled, Single and Repeated Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AUT00206 in Healthy Volunteers.
Brief Title: Safety, Blood Levels and Effects of AUT00206
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AUT011206
Record Dates: First submitted 2015-10-15; First posted 2015-10-28 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AUT00206

SUMMARY:
The study medicine is a potential future treatment for schizophrenia, an illness that affects the way that people think, feel or behave. It is not clear what causes schizophrenia, but it's been linked to chemical imbalance in the brain. It is hoped that the study medicine will activate specific sites in the brain to help correct that imbalance. Current treatments for schizophrenia don't work very well and can cause unpleasant side effects. It is hoped that the study medicine will work better, and have fewer side effects than existing medicines.

In this 2 part study (Parts A and B), the primary aim is to assess how safe the study medicine is in healthy men, aged 18-45 years, and how much of it gets into the blood. Its effects on the brain will also be tested.

In Part A, up to 24 participants will receive up to 5 single doses of the study medicine (AUT00206 or placebo) by mouth, either after fasting or after a high fat breakfast. The study medicine has never been given to humans before, so the initial doses will be small and the dose level will be increased as the study progresses. Participants may take up to 14 weeks to finish the study. They'll make up to 22 outpatient visits, and stay on the ward up to 5 times, for 3 nights in a row each time.

In Part B, 24 participants will receive daily doses of the study medicine (AUT00206 or placebo) for up to 28 days. Participants will take up to 10 weeks to finish the study. They'll make 6 outpatient visits, and stay on the ward for up to 30 nights, depending on how long we expect it to take until blood levels of the study medicine level off.

A pharmaceutical company, Autifony Therapeutics Limited, is funding the study. The study will take place at 1 centre in London.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18-45 years;
* body mass index 18.0-30.0 kg/m^2;
* in good health, as judged by medical history, medical examination, vital signs, ECG and clinical laboratory tests;
* able to communicate with study personnel; be of sufficient intelligence to understand the nature of the trial; reliable, willing, and likely to comply with the protocol;
* consent to GP being informed of their participation in the study, and to entering their details into the overvolunteering database (TOPS).

Exclusion Criteria:

* not healthy (clinically significant abnormality in screening tests, which include ECG, vital signs, physical examination, and laboratory safety tests of blood and urine);
* severe hearing impairment, or MoCA score of less than 22 points (Part B only);
* abuse of alcohol or drugs;
* taken prescription medicine during the 28 days before dosing;
* taken other medicine (except paracetamol), herbal remedies or dietary supplements during the 7 days before dosing; have had a serious reaction to any medicine, particularly medicines that work in the same way as the study medicine;
* have had any condition or operation that might affect the way the body absorbs medicines;
* have had any clinically significant disease;
* have ever attempted suicide or thought or talked about suicide, using the C-SSRS (Part B only);
* objection by GP on medical grounds;
* have donated blood, or taken part in another study, within the past 3 months; or don't agree not to donate blood, or take part in another study, during the 3 months after this study
* smoking of more than 5 cigarettes daily
* unwilling to cooperate with the requirements of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | Study duration (i.e. up to 14 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom